CLINICAL TRIAL: NCT04101175
Title: A Survey of Best Practices of Abortions at Strasbourg University Hospitals
Brief Title: Abortions at Strasbourg University Hospitals
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7472
Record Dates: First submitted 2019-07-04; First posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-07

CONDITIONS: First-trimester Pregnancy
Keywords: First-trimester pregnancy; Abortions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Request for abortion: Patient in first trimester of pregnancy in request for abortion
  Interventions: Procedure: Evaluation of the procedure of abortion

INTERVENTIONS:
Procedure: Evaluation of the procedure of abortion — Observational study using questionnaires

SUMMARY:
The number of abortions in France and Strasbourg has been stable for several years. In 2017, 1847 were performed in the Gynecology-Obstetrics Department for 6146 deliveries (23% of all pregnancies). It therefore seems important to evaluate the professional practices, but also the experiences of the patients.

ELIGIBILITY:
Inclusion criteria:

* Patient in the first trimester of pregnancy wishing an abortion
* Age: greater than or equal to 18 years.
* Patient affiliated to a social security system

Exclusion criteria:

* Patient after the first trimester pregnancy
* Patient benefiting from a legal protection measure
* Bad understanding of French.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient in the first trimester of pregnancy wishing an abortion
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Evaluate the investigator's professional practices regarding abortion, particularly in relation to the recommendations for clinical practice of the National College of French Obstetricians Gynecologists (CNGOF) published in 2016. | 6 weeks
  The patients will complete a questionnaire

SECONDARY OUTCOMES:
Evaluation of the sociological, economic and psychological factors motivating the request for abortion | 6 weeks
  The patients will complete a questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided